CLINICAL TRIAL: NCT00386399
Title: Phase II Study of Mitomycin-C in Patients With Advanced or Recurrent Pancreatic Cancer With Mutated BRCA2 Gene
Brief Title: Study of Mitomycin-C in Patients With Advanced or Recurrent Pancreatic Cancer With Mutated BRCA2 Gene
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: All consented subjects tested negative for the BRCA2 mutation, therefore, did not meet criteria to start the study, resulting in withdrawal by PI
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Van Andel Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J0626; NA_00002002 (Other: JHMIRB)
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Pancreatic Cancer
Keywords: Advanced Pancreatic Cancer; Mutated BRCA2 Gene; Recurrent Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Mitomycin

ARMS (1):
- Arm 1 (Experimental): Patients with BRCA2 gene will be treated with Mitomycin-C (MMC) on Day 1 at a dose of 10mg/m2 intravenously. This will be repeated every 28 days, which is one cycle. Treatment will continue until disease progression, serious toxicity, patient withdrawal or maximum cumulative dose of 60 mg/m2
  Interventions: Drug: Mitomycin-C

INTERVENTIONS:
Drug: Mitomycin-C — Mitomycin C, finds use as a chemotherapeutic agent by virtue of its antitumour antibiotic activity.
  Other Names: Mytomycin C

SUMMARY:
Patients will be tested for mutations in the BRCA2 gene. If they have a BRCA2 mutation, they will be treated with Mitomycin-C as described here. The patients with an identified gene mutation will also be provided with genetic counseling.

DETAILED DESCRIPTION:
Patients will be tested for mutations in the BRCA2 gene. If they have a BRCA2 mutation, they will be treated with Mitomycin-C as described here. The patients with an identified gene mutation will also be provided with genetic counseling.

Patients with BRCA2 gene will be treated with Mitomycin-C (MMC) on Day 1 at a dose of 10mg/m2 intravenously. This will be repeated every 28 days, which is one cycle. Expected adverse events and appropriate dose modifications are described in this section. Treatment will continue until disease progression, serious toxicity, patient withdrawal or maximum cumulative dose of 60 mg/m2.

Primary Objectives:

1. To determine the 6-month survival of patients with previously untreated advanced or recurrent adenocarcinoma of the pancreas with BRCA2 mutations that are treated with single agent Mitomycin-C (MMC) chemotherapy.

Secondary Objectives:

1. To determine the response rate, six-month progression free survival rate, progression-free survival and survival of patients with previously untreated advanced or recurrent adenocarcinoma of the pancreas with BRCA2 mutations who are treated with single agent MMC chemotherapy.
2. To describe the toxicity of MMC in this patient population.
3. To explore pharmacogenetic factors that may influence the toxicity and efficacy of MMC in this patient population.

ELIGIBILITY:
Inclusion Criteria

1. Histological or cytological proven adenocarcinoma of the pancreas.
2. Locally advanced unresectable or metastatic disease not amenable to curative treatment.
3. No prior treatment for advanced disease. Patient may have received adjuvant treatment after curative resection. Patients who have received gemcitabine as part of their adjuvant treatment need to have at least a 6 month progression free interval after gemcitabine has been discontinued.
4. BRCA2 deleterious mutation, or genetic variant, suspected deleterious, by DNA testing.
5. No prior treatment with MMC.
6. Age ≥18 years old.
7. ECOG PS 0-1.
8. Expected > 12 weeks survival.
9. Adequate renal, liver and bone-marrow function as determined by:
10. Ability to understand and willingness to sign a written informed consent.
11. Willingness of male and female subjects, who are not surgically sterile or post-menopausal, to use reliable methods of birth control (oral contraceptives, intrauterine devices, or barrier methods) for the duration of the study and for 30 days after the last dose of study medication.

Exclusion Criteria

1. Patients in whom histologic or cytologic diagnosis is not consistent with adenocarcinoma including adenosquamous, islet cell, cystadenoma or cystadenocarcinoma, carcinoid, small or large cell carcinoma or lymphoma.
2. Adenocarcinoma arising from a site other than pancreas (distal common bile duct, ampulla of vater or periampullary duodenum).
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
4. Patients who have had any previous surgery, excluding minor procedures, dental work, skin biopsy, etc. within 4 weeks of enrollment.
5. Uncontrolled medical conditions that could potentially increase the risk of toxicities or complications of this therapy including immunodeficiency and chronic treatment with immunosuppressors. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease.
6. Active infections.
7. History of concurrent malignancy or history of a second malignancy within the past 5 years, except squamous cell and basal cell carcinoma of the skin.
8. Participation in an investigational new drug trial within one month of starting trial.
9. Unable to provide informed consent.
10. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampin, phenobarbital or St. Johns Wort.
11. Treatment with chemotherapy within 30 days of day 1 treatment.
12. Any unresolved chronic toxicity greater than CTCAE grade 2 from previous anticancer therapy (except alopecia).
13. Pregnant women are excluded from this study because the effects of MMC on the developing fetus are not known (FDA Pregnancy Category C). Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MMC, breast feeding should be discontinued if the mother is treated with the drug.
14. Patients must not have clinically significant cardiovascular disease including myocardial infarction (within 12 months prior to randomization), unstable angina, grade II or greater peripheral vascular disease, uncontrolled congestive heart failure or uncontrolled hypertension (SBP>170, DBP>95).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
6-month overall survival | up to 6 months
  Number of participants with previously untreated advanced or recurrent adenocarcinoma of the pancreas with BRCA2 mutations that are alive after 6-months after being treated with single agent Mitomycin-C (MMC) chemotherapy.

SECONDARY OUTCOMES:
Response rate | up to 2.5 years
  Proportion of participants with reduction in tumor burden of previously untreated advanced or recurrent adenocarcinoma of the pancreas with BRCA2 mutations who are treated with single agent MMC chemotherapy.
Progression-free survival at 6 months | up to 6 months
  Number of participants who are treated with single agent MMC chemotherapy and have partial or complete response of previously untreated advanced or recurrent adenocarcinoma of the pancreas with BRCA2 mutations.
Progression-free survival | up to 2.5 years
  Number of participants who are treated with single agent MMC chemotherapy and have partial or complete response of previously untreated advanced or recurrent adenocarcinoma of the pancreas with BRCA2 mutations.
Overall survival | up to 2.5 years
  Number of participants with previously untreated advanced or recurrent adenocarcinoma of the pancreas with BRCA2 mutations who are alive after being treated with single agent MMC chemotherapy.
Toxicity as assessed by number of participants experiencing adverse events. | Up to 2.5 years
To explore pharmacogenetic factors that may influence the toxicity and efficacy of MMC in this patient population. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hidalgo, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States